CLINICAL TRIAL: NCT02331758
Title: The Influence Factors of Ovarian Response in Polycystic Ovary Syndrome Patients(PCOS) With In Vitro Fertilization and Embryo Transfer (IVF-ET) Treatment
Brief Title: The Influence Factors of Ovarian Response in PCOS Patients With IVF-ET Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing University Health Science Center (Other)
Responsible Party: Principal Investigator, Yilei He, Yilei He, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014180
Record Dates: First submitted 2014-12-31; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): The investigators use several methods to educate patients of controllable factors like lifestyle counseling, and monitor the factors like BMI and other index until the statistics become normal.
  Interventions: Behavioral: Lifestyle Counseling
- No treatment (No Intervention): Patients without any intervention and still have abnormal factors like BMI, etc.

INTERVENTIONS:
Behavioral: Lifestyle Counseling — The investigators do lifestyle counseling for PCOS patients and monitor the factors to normal level, like BMI, serum index etc.
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to explore the factors which affect ovarian response of PCOS patients with IVF-ET treatment, in order to provide predictive clinical index for the outcome of IVF-ET treatment in PCOS patients. After figuring out the controllable factors, researchers would be able to educate PCOS patients and improve the success rate while reducing the incidence of complications during the treatment at the same time.

DETAILED DESCRIPTION:
Statistics of PCOS patients like age, BMI index and others would be collected. Through distributing questionnaires and query of past cases and collecting data recorded during the ovulation process like monitoring fluctuations in blood and ultrasonic monitoring results, researchers obtain the risk factors of the occurence of Ovarian Hyperstimulation Syndrome(OHSS) in IVF-ET treatment in PCOS patients and set up an OHSS prediction model, choose controllable factors in order to make up guidance and have intervention on patients with PCOS accordingly. The investigators expect this could improve the success rate of IVF-ET treatment in patients with PCOS, provide clues and assist to reduce the risk of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PCOS
* Long schedule time of Luteal phase
* Available to trace
* Normal Prolactin level with contraceptive treatment in recent 3 months

Exclusion Criteria:

* Unwilling to participate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
oocyte number | 3 Month
  Affect the outcome of IVF-ET treatment

SECONDARY OUTCOMES:
Success Rate | 3 Month
  The success rate of IVF-ET treatment elevated
OHSS complication | 3 Month
  The number of OHSS patients reduced